CLINICAL TRIAL: NCT03047005
Title: Behavioral and Pharmacologic Treatment of Binge Eating and Obesity
Brief Title: Behavioral and Pharmacologic Treatment of Binge Eating and Obesity: Maintenance Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1506016065-M; R01DK049587 (NIH)
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Binge-Eating Disorder; Obesity
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — Naltrexone-Bupropion combination; bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NB medication (Experimental): Participants randomly assigned to this arm will receive 16 weeks of NB medication. NB medication will combine naltrexone sustained-release (SR, 32 mg/day) combined with bupropion SR (360 mg/day) taken daily in pill form.
  Interventions: Drug: NB medication (Naltrexone Bupropion combination)
- Placebo (Placebo Comparator): Participants randomly assigned to this arm will receive 16 weeks of placebo. Placebo will be inactive and taken daily in pill form.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NB medication (Naltrexone Bupropion combination) — NB medication
  Other Names: Contrave
  Arms: NB medication
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will test the effectiveness and relative efficacy of naltrexone/bupropion medication as a maintenance therapy for the treatment of binge eating disorder (BED) in patients with obesity. This is a controlled test of whether, amongst responders to acute treatments, naltrexone/bupropion medication results in superior maintenance and longer-term outcomes compared with placebo.

DETAILED DESCRIPTION:
Binge eating disorder (BED), the most prevalent formal eating disorder, is associated strongly with obesity and bio-psychosocial impairment. Improved treatments for patients with obesity and BED are needed that can produce sustained clinical outcomes and promote weight loss. This study (maintenance stage) RCT will provide new and novel findings from a controlled test, amongst responders to acute treatments, whether NB medication results in superior maintenance and longer-term outcomes than placebo. This is the first controlled test of maintenance pharmacotherapy for BED and will be only the third RCT for BED of any medication with follow-up after medication discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Participated in acute treatment for binge-eating disorder and obesity;
* Had a positive response to acute treatment;
* Available for the duration of the treatment and follow-up (20 months);
* Read, comprehend, and write English at a sufficient level to complete study-related materials; and
* Able to travel to study location (New Haven, CT) for monthly visits.

Exclusion Criteria:

* Currently taking anti-depressant medications;
* Currently taking opioid pain medications or drugs;
* Currently taking medications that influence eating/weight;
* History of seizures;
* Current substance use disorder or other severe psychiatric disturbance (e.g., suicidality);
* Past or current anorexia nervosa, bulimia nervosa;
* Pregnant or breastfeeding;
* Medical status judged by study physician as contraindication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Grilo, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The main study (acute treatment results) can be found in NCT03045341. Two participants dropped prior to beginning the medication.
Period: Overall Study
Arm/Group | NB Medication | Placebo
Started | 32 | 34
Completed | 29 | 28
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NB Medication | Placebo | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.40 (11.70) | 43.60 (11.80) | 46.92 (12.15)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Men | 3 | 6 | 9
  Women | 28 | 28 | 56
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 29 | 28 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 25 | 22 | 47
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Binge Eating Frequency (Continuous)
Description: Binge eating will be assessed by interview and self-report and the primary outcome is frequency. Frequency will be defined continuously (analyzed dimensionally).
Time Frame: Post-treatment (4 months)
Measure: Mean (Standard Deviation); unit: binge eating days per month
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 29 | 28
binge eating days per month | 0.86 (2.15) | 3.25 (7.06)
Statistical Analysis 1: Comparison: NB Medication vs Placebo; Test type: Superiority — Analyses used all available data. Analyses to compare treatments were all intent-to-treat; p = .07, Mixed Models Analysis; Analyses were performed for all randomized patients who attended the first treatment session. Model adjusted for stage 1 treatment condition

2. Primary Outcome: Change in Body Mass Index
Description: BMI is calculated using measured height and weight. We report percent change in weight from baseline. Negative values indicate weight loss.
Time Frame: baseline and Post-treatment (4 months)
Measure: Mean (Standard Deviation); unit: percentage weight change
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 29 | 26
percentage weight change | -0.03 (.05) | .01 (.04)
Statistical Analysis 1: Comparison: NB Medication vs Placebo; Test type: Superiority — Analyses used all available data. Analyses to compare treatments were all intent-to-treat; p = .01, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Binge Eating Frequency (Continuous)
Description: as for outcome 1
Time Frame: 6-Month Follow-up
Measure: Mean (Standard Deviation); unit: eating events/28 days
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 23 | 21
eating events/28 days | 1.57 (4.42) | 2.43 (4.92)

4. Secondary Outcome: Binge Eating Frequency (Continuous)
Description: as for outcome 1
Time Frame: 12-Month Follow-up
Measure: Mean (Standard Deviation); unit: eating events/28 days
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 17 | 22
eating events/28 days | 3.35 (6.58) | 2.77 (6.15)

5. Secondary Outcome: Change in Body Mass Index (BMI)
Description: BMI is calculated using measured height and weight. We report percent change in BMI from baseline. Negative values indicate weight loss.
Time Frame: Baseline to 6-Month Follow-up
Measure: Mean (Standard Deviation); unit: percentage change in BMI
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 23 | 21
percentage change in BMI | .004 (.065) | .026 (.063)

6. Secondary Outcome: Change in Body Mass Index
Description: as for outcome 5
Time Frame: Baseline to 12-Month Follow-up
Measure: Mean (Standard Deviation); unit: percentage change in BMI
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 16 | 22
percentage change in BMI | .025 (.079) | .042 (.076)

ADVERSE EVENTS:
Time Frame: Month 1
Description: Participants were interviewed by research clinicians. For non-serious adverse events that were listed as >5% on the package insert for "Contrave" (naltrexone HCl/ bupropion HCl), we provide the total participants [all available data] who reported the adverse event at month 1. For serious adverse events, we provide the total participants [all available data] who reported the adverse event over the course of the study.
Arm/Group | NB Medication | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34
Other Adverse Events (participants affected / at risk) | 21/32 | 18/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NB Medication (N=32) | Placebo (N=34)
Hypertensive Crisis (Cardiac disorders) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NB Medication (N=32) | Placebo (N=34)
Constipation (Gastrointestinal disorders) | 10 | 5
Diarrhea (Gastrointestinal disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 8 | 3
Vomiting (Gastrointestinal disorders) | 3 | 3
Dizziness (General disorders) | 4 | 4
Dry Mouth (General disorders) | 10 | 3
Headache (General disorders) | 9 | 4
Insomnia (General disorders) | 7 | 9
Anxiety (Psychiatric disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT03047005/Prot_SAP_000.pdf